CLINICAL TRIAL: NCT03117283
Title: Laparoscopic Total Gastrectomy With Bursectomy in a Left Outside Bursa Omentalis Approach Versus Laparoscopic Total Gastrectomy Without Bursectomy for Advanced Posterior Gastric Wall Cancer: a Randomized Controlled Study
Brief Title: Laparoscopic Total Gastrectomy With Versus Without Bursectomy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Wei Wang, Wei Wang M.D., PhD., Guangdong Provincial Hospital of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GDPHCM-GI-02
Record Dates: First submitted 2017-04-07; First posted 2017-04-17 (Actual); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: Laparoscopic Gastrectomy; Laparoscopic Bursectomy; A Left Outside Bursa Omentalis Approach
Keywords: Laparoscopic surgery; Radical total gastrectomy; Bursectomy; Advanced posterior gastric wall cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LTG with Bursectomy (Experimental): laparoscopic D2 radical total gastrectomy with bursectomy using a left outside bursa omentalis approach
  Interventions: Procedure: Laparoscopic D2 radical total gastrectomy with bursectomy using a left outside bursa omentalis approach
- LTG without Bursectomy (Sham Comparator): laparoscopic D2 radical total gastrectomy without bursectomy
  Interventions: Procedure: Laparoscopic D2 radical total gastrectomy without bursectomy

INTERVENTIONS:
Procedure: Laparoscopic D2 radical total gastrectomy with bursectomy using a left outside bursa omentalis approach — Patients with advanced posterior gastric wall cancer including in the laparoscopic total gastrectomy (LTG) with bursectomy group will undergo laparoscopic D2 radical total gastrectomy with bursectomy using a left outside bursa omentalis approach.
  Arms: LTG with Bursectomy
Procedure: Laparoscopic D2 radical total gastrectomy without bursectomy — Patients who are included in the laparoscopic total gastrectomy (LTG) without bursectomy group will undergo laparoscopic D2 radical total gastrectomy without bursectomy in a conventional manner.
  Arms: LTG without Bursectomy

SUMMARY:
Bursectomy is widely performed in open surgery for advanced gastric cancer in East Asia. However laparoscopic D2 radical total gastrectomy with complete bursectomy is difficult and rare performed. Herein, we conduct a single-centre randomized controlled trial to explore the safety and feasibility of totally laparoscopic D2 radical total gastrectomy using a left outside bursa omentalis approach for achieving complete bursectomy.

DETAILED DESCRIPTION:
Although, the clinical value of bursectomy in addition to D2 lymphadenectomy in radical gastrectomy for curable gastric cancer is controversial. Data analysis of the nationwide registry of gastric cancer in Japanese revealed that 10.7% of patients with subserosal and serosal positive cancer developed peritoneal recurrence after radical gastrectomy. Some trials, although, indicated a biologically reasonable but statistically non-significant advantage to bursectomy. But for patients with posterior gastric wall trans-serosal disease, such micrometastases can constitute the seeds of later recurrence. The non-bursectomy showed worse overall survival. Early removal of micrometastases and cancer cells deposited might prove beneficial and a possible therapeutic effect. In any case, the authors reasonably concluded that bursectomy should not be abandoned at this time. The hypothesis that it might actually enhance survival should be entertained. In the past decades, Japanese, Korea, Chinese and even Turkey, surgeons have continued to performed bursectomy and lymph nodes dissection as the conventional open procedures for advanced gastric cancer. Lymph nodes dissection and bursectomy is routinely regarded as a standard surgical procedure during radical open gastrectomy for tumors penetrating the serosa of the posterior gastric wall. Complete bursectomy and lymphadenectomy in open radical gastrectomy may represents a formidable challenge to the best of surgeons and its influences on operative morbidity and mortality, but it can be also safely performed in high volume experience centers or by experienced surgeons with mortality rate of <1% and morbidity rates around 14%.

Generally speaking, bursectomy is incomplete without total gastrectomy. The concept of bursectomy mentioned above is always almost confined to removal of the local anterior membrane of the transverse mesocolon and pancreatic capsule and to open radical gastrectomy. With the generalization and development of laparoscopic technology, laparoscopic surgery for advanced gastric cancer as clinical study has extensively performed in Asia.The investigators take the lead in carrying out laparoscopic bursectomy and D2 radical gastrectomy by. Herein, the investigators conduct a single-centre randomized controlled trial to explore the safety and feasibility of totally laparoscopic D2 radical total gastrectomy using a left outside bursa omentalis approach for achieving complete bursectomy.

ELIGIBILITY:
Inclusion Criteria:

* Primary gastric adenocarcinoma diagnosed pathologically by endoscopic biopsy
* Tumor located in the posterior wall of upper and middle third stomach estimated by endoscopy and CT scan
* Informed consent
* Eastern Cooperative Oncology Group (ECOG): 0 ot 1
* American Society of Anesthesiologists （ASA） score: Ⅰto Ⅲ

Exclusion Criteria:

* Pregnancy or female in suckling period
* Contraindication to general anesthesia (severe cardiac and/or pulmonary disease)
* Severe mental disease
* Emergency operation due to complication (bleeding, perforation or obstruction) caused by primary tumor

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2017-03-28 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Early morbidity | 30 days
  The early morbidity is defined as the adverse event observed during peri-operative time.

SECONDARY OUTCOMES:
Operative time | Intraoperative
  The mean operative time of the procedures
Lymph node | 14 days
  This outcome consists of the number of total lymph nodes harvested and the number of lymph nodes in the wall of bursa omentalis
First ambulation | 30 days
  The time to first ambulation
3-year survival | 3 years
  3-year disease free survival rate
5-year survival | 5 years
  5-year overall survival rate
Estimated blood loss | Intraoperative
  The mean estimated blood loss
First flatus | 30 days
  The time to first flatus
First liquid diet | 30 days
  The time to liquid diet
Hospital stay | 30 days
  Postoperative hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine; Wenjun Xiong, Principal Investigator — Guangdong Provincial Hospital of Traditional Chinese Medicine
Locations (1):
- Guangdong Province Hospital of Chinese Medicine, the Second Affiliated Hospital of Guangzhou University of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
The data has not been published.

REFERENCES:
- [Result] Hundahl SA. The potential value of bursectomy in operations for trans-serosal gastric adenocarcinoma. Gastric Cancer. 2012 Jan;15(1):3-4. doi: 10.1007/s10120-011-0121-6. No abstract available. PMID 22160297
- [Result] Japanese Gastric Cancer Association Registration Committee; Maruyama K, Kaminishi M, Hayashi K, Isobe Y, Honda I, Katai H, Arai K, Kodera Y, Nashimoto A. Gastric cancer treated in 1991 in Japan: data analysis of nationwide registry. Gastric Cancer. 2006;9(2):51-66. doi: 10.1007/s10120-006-0370-y. PMID 16767357
- [Result] Fujita J, Kurokawa Y, Sugimoto T, Miyashiro I, Iijima S, Kimura Y, Takiguchi S, Fujiwara Y, Mori M, Doki Y. Survival benefit of bursectomy in patients with resectable gastric cancer: interim analysis results of a randomized controlled trial. Gastric Cancer. 2012 Jan;15(1):42-8. doi: 10.1007/s10120-011-0058-9. Epub 2011 May 15. PMID 21573917
- [Result] Imamura H, Kurokawa Y, Kawada J, Tsujinaka T, Takiguchi S, Fujiwara Y, Mori M, Doki Y. Influence of bursectomy on operative morbidity and mortality after radical gastrectomy for gastric cancer: results of a randomized controlled trial. World J Surg. 2011 Mar;35(3):625-30. doi: 10.1007/s00268-010-0914-5. PMID 21161652
- [Result] Kayaalp C, Piskin T, Olmez A. Complications of bursectomy after radical gastrectomy for gastric cancer. World J Surg. 2012 Jan;36(1):229; author reply 230. doi: 10.1007/s00268-011-1218-0. No abstract available. PMID 21833663
- [Result] Hirao M, Kurokawa Y, Fujita J, Imamura H, Fujiwara Y, Kimura Y, Takiguchi S, Mori M, Doki Y; Osaka University Clinical Research Group for Gastroenterological Study. Long-term outcomes after prophylactic bursectomy in patients with resectable gastric cancer: Final analysis of a multicenter randomized controlled trial. Surgery. 2015 Jun;157(6):1099-105. doi: 10.1016/j.surg.2014.12.024. Epub 2015 Feb 20. PMID 25704429
- [Result] Wang W, Xiong W, Liu Z, Luo L, Zheng Y, Tan P, Diao D, Zou L, Wan J. Clinical significance of No. 10 and 11 lymph nodes posterior to the splenic vessel in D2 radical total gastrectomy: An observational study. Medicine (Baltimore). 2016 Aug;95(32):e4581. doi: 10.1097/MD.0000000000004581. PMID 27512888
- [Result] Wang W, Liu Z, Xiong W, Zheng Y, Luo L, Diao D, Wan J. Totally laparoscopic spleen-preserving splenic hilum lymph nodes dissection in radical total gastrectomy: an omnibearing method. Surg Endosc. 2016 May;30(5):2030-5. doi: 10.1007/s00464-015-4438-9. Epub 2015 Jul 23. PMID 26201417